CLINICAL TRIAL: NCT01973257
Title: Perfusion and Diffusion Mechanism of Intervertebral Disc-Significance With Age, Degeneration, Posture and Stress Loading.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 200612091R
Record Dates: First submitted 2013-10-24; First posted 2013-10-31 (Estimated); Last update posted 2013-11-01 (Estimated); Status verified 2013-10

CONDITIONS: Spinal Cord Injury, Degenerative Spinal Disease.
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Who Masked: Participant

ARMS (1):
- select from the option menu (Experimental): select from the option menu
  Interventions: Procedure: imaging diagnostics

INTERVENTIONS:
Procedure: imaging diagnostics

SUMMARY:
The purpose of our study is to evaluate the perfusion of the IVDs and their diffusion ability by using the Dynamic contrast-enhanced MR perfusion technique and Diffusion weighted image with ADC value measurement, and to determine the relationship between these data and the degeneration of IVDs, the different posture, and different stress-loading status.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a diagnosis of spinal cord injury and degenerative spinal disease
* Normal volunteers

Exclusion Criteria:

- Patients with cancer and infection.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2007-08; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
Disc Perfusion | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Tiffany Ting-Fang Shih, Principal Investigator — Department of Medical Image, National Taiwan University Hospital
Locations (1):
- Tiffany Ting-Fang Shih, Taipei, Taiwan